CLINICAL TRIAL: NCT01394900
Title: Couples-Based HIV/STI Prevention for Drug-Involved, Black MSM
Brief Title: Connect 'n Unite: Couples-Based HIV/STI Prevention for Drug-Involved, Black MSM
Acronym: CNU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AAAI5452; 1R01DA030296-01A1 (NIH)
Record Dates: First submitted 2011-07-13; First posted 2011-07-15 (Estimated); Last update posted 2024-06-04 (Actual); Status verified 2024-06

CONDITIONS: HIV; Sexually Transmitted Infections
Keywords: HIV; sexually transmitted infection; STI; men who have sex with men; MSM; couples; African American; Black
MeSH Terms: conditions — Sexually Transmitted Diseases; Homosexuality | interventions — 1-(2-chloroethyl)-1-nitrosourea; Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- CNU intervention (Experimental): African American/Black men who have sex with men (MSM) in same sex intimate relationships in which at least one partner is illicitly using psychostimulants and/or psychoactive substances will receive 4 sessions of CNU intervention
  Interventions: Behavioral: CNU Intervention
- WP intervention (Active Comparator): African American/Black men who have sex with men (MSM) in same sex intimate relationships in which at least one partner is illicitly using psychostimulants and/or psychoactive substances will receive 4 sessions of general wellness promotion (WP) intervention
  Interventions: Behavioral: WP Intervention

INTERVENTIONS:
Behavioral: CNU Intervention — Notions that strengthen the closeness with one's partner, connect with similar couples, and visibly strengthen a community as key to combating dynamics that cause poor communication, isolation, fragmentation of the Black MSM community.
  Other Names: Connect 'n Unite (CNU) Intervention
  Arms: CNU intervention
Behavioral: WP Intervention — Attention control condition - WP focuses on nutrition, fitness, healthcare, and stress management. Given the prevalence of health problems among the target population, WP emphasizes adherence to medical guidance and medication regimens.
  Other Names: Wellness Promotion (WP) Intervention
  Arms: WP intervention

SUMMARY:
The study has the following primary aims: (1) to test whether participants assigned to CNU (a 7-session, manualized intervention entitled "Connect 'n Unite") engage in lower HIV/STI behavioral risk compared to participants assigned to WP (a wellness promotion attention control condition); (2) to test whether participants assigned to CNU have lower cumulative incidence of STIs-chlamydia and gonorrhea-confirmed via biological assay compared to participants assigned to WP; and (3) to test whether participants assigned to CNU engage in less drug use compared to participants assigned to WP.

DETAILED DESCRIPTION:
This study addresses the overrepresentation of the African American/Black community among those living with HIV/AIDS in the U.S. as well as men who have sex with men (MSM), the transmission category that accounts for the majority of HIV infections. In the absence of a vaccine or cure for HIV infection, behavioral risk reduction represents the best public health tool for prevention of HIV transmission. The proposed randomized clinical trial will rigorously test an innovative, couples-based intervention targeting the intersection of stimulant use and sexual risk behavior among racial/ethnic and sexual minorities, with the ultimate goal providing an evidence-based intervention that can be delivered in drug treatment and other service settings to reduce the spread of HIV among stimulant-using, African American/Black MSM.

ELIGIBILITY:
Inclusion Criteria:

* Male
* At least 18 years old
* Report having a "primary/main male partner" operationalized as a male with whom he has had an ongoing sexual relationship over the prior 6 months and has an emotional bond with more than any person
* Self-identify as African American and/or Black, or identify having a main partner who self-identifies in this manner
* Report using a illicit use of psychostimulant and/or psychoactive drugs in the past 90 days (or has a main male partner who meets this criterion)
* Report having unprotected anal sex with a man who is a non-main partner in the past 90 days (or has a main male partner who meets this criterion)
* Identify each other as their main partner

Exclusion Criteria:

* Either partner reports the occurrence of ≥1 incident of severe intimate partner violence (IPV) within the relationship in the past year as assessed using the Revised Conflict Tactics Scales
* Either partner has a language or cognitive impairment that prevents comprehension of study procedures as assessed during informed consent
* Either partner reports being currently involved (i.e., has not completed the final follow-up assessment) in an HIV prevention research study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 424 (Actual)
Dates: Start 2012-07; Primary Completion 2016-12-31 (Actual); Study Completion 2019-08-02 (Actual)

PRIMARY OUTCOMES:
Difference in number of unprotected acts of anal intercourse between 2 groups | 12 months
  To test whether participants assigned to the CNU intervention engage in lower HIV/STI behavioral risk compared to participants assigned to the WP attention control condition using the following primary outcome - number of unprotected acts of anal intercourse.

SECONDARY OUTCOMES:
Difference in incidence of sexually transmitted infections (STIs) between 2 groups | 12 months
  To test whether participants assigned to CNU have lower cumulative incidence of STIs confirmed via biological assay compared to participants assigned to WP.
Difference in number of illicit drug use between 2 groups | 12 months
  To test whether participants assigned to CNU engage in less drug use compared to participants assigned to WP.

CONTACTS AND LOCATIONS:
Overall Officials: Elwin Wu, PhD, Principal Investigator — Columbia University
Locations (1):
- Columbia University School of Social Work, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided